CLINICAL TRIAL: NCT00182715
Title: A Three-Arm Randomised Controlled Trial Comparing Either Continuous Chemotherapy Plus Cetuximab or Intermittent Chemotherapy With Standard Continuous Palliative Combination Chemotherapy With Oxaliplatin and a Fluoropyrimidine in First Line Treatment of Metastatic Colorectal Cancer (COIN)
Brief Title: Combination Chemotherapy With or Without Cetuximab as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Velindre NHS Trust (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000440085; UKM-MRC-COIN-CR10; EU-20516; EUDRACT-2004-002951-16; ISRCTN27286448
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage IV colon cancer; adenocarcinoma of the rectum; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether combination chemotherapy and cetuximab are more effective than combination chemotherapy alone in treating colorectal cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and cetuximab to see how well they work compared to combination chemotherapy alone as first-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with metastatic colorectal adenocarcinoma treated with continuous combination chemotherapy comprising oxaliplatin, leucovorin calcium, and fluorouracil (OxMdG) or oxaliplatin and capecitabine (XELOX) with vs without cetuximab vs intermittent combination chemotherapy with OxMdG or XELOX as first-line therapy.

Secondary

* Compare time of disease control and progression- and failure-free survival of patients treated with these regimens.
* Compare response in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the cost effectiveness of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a multicenter, open label, randomized, controlled study. Patients are randomized to 1 of 3 treatment arms.

* Arm I (continuous chemotherapy): Patients receive 1 of the following combination chemotherapy regimens of their choice (or as per participating center):

  * OxMdG: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  * XELOX: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II (continuous chemotherapy and cetuximab): Patients receive OxMdG or XELOX as in arm I. Patients also receive cetuximab IV over 1-2 hours on days 1 and 8 (for patients receiving OxMdG) OR days 1, 8, and 15 (for patients receiving XELOX). Treatment with OxMdG and cetuximab repeats every 14 days in the absence of disease progression or unacceptable toxicity. Treatment with XELOX and cetuximab repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm III (intermittent chemotherapy): Patients receive OxMdG or XELOX as in arm I. Treatment with OxMdG repeats every 14 days for up to 6 courses (12 weeks). Treatment with XELOX repeats every 21 days for up to 4 courses (12 weeks). Patients with disease progression after 12 weeks of therapy are removed from study treatment. Patients with stable or responding disease after 12 weeks of therapy stop treatment and undergo clinical evaluation at least every 6 weeks (treatment break) until disease progression or clinical deterioration. Upon evidence of disease progression or clinical deterioration, patients restart treatment with OxMdG or XELOX as before and continue to alternate 12 weeks of treatment with treatment breaks in the absence of disease progression or unacceptable toxicity Quality of life is assessed at baseline, 6 weeks, 12 weeks, and then every 12 weeks thereafter.

After completion of study treatment, patients are followed every 12 weeks for survival.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2,421 patients (807 per treatment arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma, defined by 1 of the following:

  * Histologically confirmed primary adenocarcinoma of the colon or rectum with clinical or radiological evidence of advanced and/or metastatic disease
  * Histologically or cytologically confirmed metastatic adenocarcinoma with clinical or radiological evidence of primary colorectal tumor
* Unidimensionally measurable disease
* Inoperable metastatic or locoregional disease

  * Ineligible for hepatic resection after first-line combination chemotherapy
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* AST or ALT ≤ 2.5 times ULN

Renal

* Creatinine clearance or glomerular filtration rate ≥ 50 mL/min

Cardiovascular

* No poorly controlled angina
* No myocardial infarction within the past 3 months

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be considered fit to undergo combination chemotherapy
* No psychiatric or neurological condition that would preclude study compliance or giving informed consent
* No partial or complete bowel obstruction
* No other malignant disease that would preclude study treatment
* No preexisting neuropathy > grade 1
* No known hypersensitivity reaction to any of the components of study drugs
* No known DPD deficiency or personal or family history suggestiv of DPD deficiency
* No other severe uncontrolled medical illness that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic palliative chemotherapy for metastatic disease
* No prior oxaliplatin
* More than 1 month since prior adjuvant fluorouracil (5-FU) (with or without leucovorin calcium), capecitabine, or irinotecan
* More than 1 month since prior rectal chemoradiotherapy with 5-FU (with or without leucovorin calcium) or capecitabine

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy

Surgery

* Not specified

Other

* No concurrent brivudine or sorivudine (for patients receiving capecitabine on study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2421 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 2 years

SECONDARY OUTCOMES:
Progression-free survival at 2 years
Failure-free survival at 2 years
Response by RECIST criteria at 12 and 24 weeks
Toxicity by NCI Common Toxicity Criteria version 3 throughout treatment and at follow-up
Time of disease control at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Maughan, MD, Study Chair — Velindre NHS Trust
Locations (82):
- Ireland (10):
  - Mercy University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford
- United Kingdom (72):
  - North Hampshire Hospital, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital NHS Trust, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dorset County Hospital, Dorchester, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Princess Alexandra Hospital, Essex, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - Cookridge Hospital, Leeds, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - University College of London Hospitals, London, England
  - Royal Free and University College Medical School, London, England
  - Queen Elizabeth Hospital - Woolwich, London, England
  - Cancer Research UK Clinical Groups at Guy's King's & St. Thomas' Hospitals, London, England
  - St. George's Hospital, London, England
  - Royal Marsden - London, London, England
  - Hammersmith Hospital, London, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Southport and Formby District General Hospital, Merseyside, England
  - St. Mary's Hospital, Newport, England
  - North Tyneside Hospital, North Shields, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Poole Hospital NHS Trust, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Whiston Hospital, Prescot Merseyside, England
  - Royal Preston Hospital, Preston, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Salisbury District Hospital, Salisbury, England
  - Scarborough General Hospital, Scarborough, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton General Hospital, Southampton, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Sunderland Royal Hospital, Sunderland, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Walsall Manor Hospital, Walsall, England
  - Good Hope Hospital Trust, West Midlands, England
  - Royal Hampshire County Hospital, Winchester, England
  - Worcester Royal Hospital, Worcester, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales

REFERENCES:
- [Result] Adams RA, Meade AM, Seymour MT, Wilson RH, Madi A, Fisher D, Kenny SL, Kay E, Hodgkinson E, Pope M, Rogers P, Wasan H, Falk S, Gollins S, Hickish T, Bessell EM, Propper D, Kennedy MJ, Kaplan R, Maughan TS; MRC COIN Trial Investigators. Intermittent versus continuous oxaliplatin and fluoropyrimidine combination chemotherapy for first-line treatment of advanced colorectal cancer: results of the randomised phase 3 MRC COIN trial. Lancet Oncol. 2011 Jul;12(7):642-53. doi: 10.1016/S1470-2045(11)70102-4. Epub 2011 Jun 5. PMID 21641867
- [Result] Maughan TS, Adams RA, Smith CG, Meade AM, Seymour MT, Wilson RH, Idziaszczyk S, Harris R, Fisher D, Kenny SL, Kay E, Mitchell JK, Madi A, Jasani B, James MD, Bridgewater J, Kennedy MJ, Claes B, Lambrechts D, Kaplan R, Cheadle JP; MRC COIN Trial Investigators. Addition of cetuximab to oxaliplatin-based first-line combination chemotherapy for treatment of advanced colorectal cancer: results of the randomised phase 3 MRC COIN trial. Lancet. 2011 Jun 18;377(9783):2103-14. doi: 10.1016/S0140-6736(11)60613-2. Epub 2011 Jun 5. PMID 21641636
- [Result] Adams RA, Meade AM, Madi A, Fisher D, Kay E, Kenny S, Kaplan RS, Maughan TS. Toxicity associated with combination oxaliplatin plus fluoropyrimidine with or without cetuximab in the MRC COIN trial experience. Br J Cancer. 2009 Jan 27;100(2):251-8. doi: 10.1038/sj.bjc.6604877. PMID 19165196
- [Result] Maughan T: Cetuximab (C), oxaliplatin (Ox) and fluoropyrimidine (Fp): toxicity during the first 12 weeks of treatment for the first 804 patients entered into the MRC COIN (CR10) trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-4070, 2007.